CLINICAL TRIAL: NCT03549468
Title: The Effect of Low LEVel TrAgus STimulation on the Electrophysiological Substrate of Patients With Ischemic CardioMyopathy
Brief Title: The Effect of Low LEVel TrAgus STimulation on the Electrophysiological Substrate of Patients With Ischemic CardioMyopathy Substrate of Subjects With Ischemic CardioMyopathy
Acronym: ELEVATE-ICM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8672
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Ischemic Cardiomyopathy
Keywords: ischemic cardiomyopathy; neuromodulation; repolarization alternans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- low level tragus stimulation (LLTS) (Experimental): Patients with ischemic cardiomyopathy (left ventricular ejection fraction <35%) and heart failure who already have an implantable device with an atrial lead (dual chamber defibrillator or biventricular defibrillator) will undergo sequentially 1. Sham LLTS (5min), 2. Active LLTS at 5Hz (15min) and 20Hz (15min) and 3. Active LLTS group with atrial pacing at 100bpm at 5Hz (15min) and 20Hz (15min).
  Interventions: Device: Low level tragus stimulation

INTERVENTIONS:
Device: Low level tragus stimulation — All patients will undergo sequentially: sham stimulation; LLTS (5Hz), LLTS (20Hz). The sequence will be repeated during atrial pacing at 100bpm

SUMMARY:
Patients with ischemic cardiomyopathy (left ventricular ejection fraction <35%) and heart failure who already have an implantable device with an atrial lead (dual chamber defibrillator or biventricular defibrillator) will undergo sequentially 1. Sham low level tragus stimulation (LLTS) (5min), 2. Active LLTS at 5Hz (15min) and 20Hz (15min) and 3. Active LLTS group with atrial pacing at 100bpm at 5Hz (15min) and 20Hz (15min). The latter is required to examine the effect of LLTS on RA independent of heart rate. Repolarization alternans will be measured by analyzing a regular 12-lead ECG using a custom-made software.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic cardiomyopathy (LVEF <35%) and heart failure
2. Implantable device with an atrial lead (dual chamber ICD or CRT-D)
3. Sinus rhythm at the time of the study

Exclusion Criteria:

1. Recent (<6 months) stroke or myocardial infarction
2. Persistent atrial fibrillation
3. Recurrent vaso-vagal syncopal episodes
4. Unilateral or bilateral vagotomy
5. Pregnancy or breast feeding
6. Uncontrolled diabetes or hypertension
7. Sick sinus syndrome and 2nd or 3rd degree AV block (without a pacemaker)
8. Bifascicular block or prolonged first degree block
9. Hypotension due to autonomic dysfunction
10. Inability or unwillingness to understand and/or sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Repolarization alternans, an ECG measure for susceptibility to VT/VF | during acute stimulation procedure
  Repolarization alternans will be measured by analyzing a regular 12-lead ECG using a custom-made software

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States